CLINICAL TRIAL: NCT05768568
Title: Comparison of Plaque Removal Efficacy of Powered and Manual Toothbrush Among Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mohsin Haider, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MH21
Record Dates: First submitted 2021-09-05; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy, Mixed
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: CP children who will meet the inclusion criteria will be assigned into two groups. Baseline debris, calculus and gingival and plaque status will be recorded using Oral Hygiene Index Simplified (OHI-S) and gingival & plaque index (PI, GI). The group I will receive a conventional manual toothbrush and group II will be given powered toothbrush. After 4 weeks will receive powered brush and group II will receive manual brush. After 4 weeks again the subjects will be assessed again for PI, GI, OHI-S. The scores will be compared and analyzed from baseline, after first phase and after second phase of interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Manual Toothbrush.
  Interventions: Device: Manual Toothbrush and Powered Toothbrush
- Group II (Active Comparator): Powered Toothbrush
  Interventions: Device: Manual Toothbrush and Powered Toothbrush

INTERVENTIONS:
Device: Manual Toothbrush and Powered Toothbrush — Manual Toothbrush will be mechanically (hand) driven Powered Toothbrush will be battery operated

SUMMARY:
CHildren of Cerebral Palsy(CP) are at high risk of developing dental diseases most commonly periodontitis and caries. Neuromuscular and psychological impact makes it difficult for the CP child to clean dental plaque from the surface of the teeth.inability to perform coordinated movements too makes brushing very difficult and hence it worsens the oral hygiene status.

Hence the objective of the study is to assess plaque removal efficacy of powered toothbrush versus manual toothbrush evaluated by improvement in oral hygiene status of patients with Cerebral Palsy CP children who meet inclusion exclusion criteria will be assessed at different time intervals via Oral hygiene index simplified (OHI-S), plaque index (PI) and gingival index (GI) Scores will be compared and analyzed from baseline, after first phase and after second phase of interventions.

DETAILED DESCRIPTION:
Children with cerebral palsy manifests neurologically associated muscular dysfunction. They face difficulty in maintaining posture, gait and locomotion, leading to restricted movements. They are at a higher risk of developing dental diseases most commonly periodontitis and caries. Neuromuscular and psychological impact makes it difficult for the CP child to clean dental plaque from the surface of the teeth. The main cause of dental diseases in CP is ineffective removal of dental plaque. This is due to lack of motor and neuromuscular dysfunction with an inability to understand and comprehend oral hygiene instructions and unable to carryout well-coordinated movements for instance tooth brushing. In a disadvantaged population interventions should be introduced at an early phase of life encouraging it to become part of CP child's daily oral hygiene maintenance regime.

Hence the objective of the study was designed to assess plaque removal efficacy of powered toothbrush versus manual toothbrush evaluated by improvement in oral hygiene status of patients with Cerebral Palsy CP children who will meet the inclusion criteria will be assigned into two groups. Baseline debris, calculus and gingival and plaque status will be recorded using Oral Hygiene Index Simplified (OHI-S) and gingival & plaque index (PI, GI). The group I will receive a conventional manual toothbrush and group II will be given powered toothbrush. After 4 weeks,will receive powered brush and group II will receive manual brush. After 4 weeks again the subjects will be assessed again for PI, GI, OHI-S. The scores will be compared and analyzed from baseline, after first phase and after second phase of interventions. Repeated measures two way ANOVA with Post Hoc Tukey test. Repeated measures two way ANOVA with Post Hoc Tukey test will be applied on mean GI, PI and OHI-S. Results of phase-I and phase-II will be compared and analyzed

ELIGIBILITY:
Inclusion Criteria:

1. CP Children aged 12-15 years
2. CP children with OHI-S score >1.3 and GI score >1 & PI score >1
3. Subjects with positive consent from schools and parents
4. Presence of at least 20 teeth in the mouth
5. Independent (mild) CP patients - who are able to perform tooth brushing under supervision assessed by caregiver's account of daily activities.
6. Mentally stable

Exclusion Criteria:

1. Inability to cooperate with the oral examination
2. Severe neuromuscular incoordination
3. Reluctant or Unable to comprehend consent /or withdrawal of consent
4. Participant with calculus deposits at baseline
5. Lack of Manual dexterity to perform oral hygiene
6. Underlying systemic disease
7. Participant requiring emergency dental treatment

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Oral Hygiene Status assessed by Oral Hygiene Index Simplified (OHI-S) | 3 months
  According to this Oral Hygiene Index Simplified (OHI-S) The oral hygiene status will be classified as Good (0-1.2), Fair (1.3-3.0), Poor (3.1-6.0)
Oral Hygiene Status assessed by Gingival Index (GI) | 3 months
  Gingival status will be classified as Mild (0.1-1), Moderate (1.1-2) and Sever (2.1-3)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Haider, BDS, Principal Investigator — Dow University
Locations (1):
- Al Umeed Rehabilitation Association (AURA), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No